CLINICAL TRIAL: NCT00045266
Title: An Open-Label, Long Term, Safety, and Tolerability Study of VEGF Trap in Patients With Incurable, Relapsed or Refractory Solid Tumors or Lymphoma
Brief Title: VEGF Trap in Treating Patients With Solid Tumors or Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: REGENERON-VGF-ST-0105; MSKCC-02020; CDR0000256462 (Registry Identifier: PDQ (Physician Data Query)); NCI-G-02-2101
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; unspecified adult solid tumor, protocol specific; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — aflibercept

INTERVENTIONS:
Biological: ziv-aflibercept

SUMMARY:
RATIONALE: VEGF Trap may stop the growth of solid tumors or non-Hodgkin's lymphoma by stopping blood flow to the cancer.

PURPOSE: Phase I trial to study the effectiveness of VEGF Trap in treating patients who have relapsed or refractory solid tumors or non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the long-term safety and tolerability of VEGF Trap in patients with incurable relapsed or refractory solid tumors or non-Hodgkin's lymphoma with stable or responding disease after receiving treatment on protocol MSKCC-01131.
* Determine the biological effect of this therapy on suppressing tumor growth or progression in these patients.
* Determine the steady state concentration of VEGF Trap over time in these patients.
* Determine whether patients develop antibodies to this therapy during extended exposure.

OUTLINE: This is an extension study for patients who showed evidence of stable disease or complete or partial remission after completing treatment on protocol MSKCC-01131.

Patients continue to receive VEGF Trap subcutaneously once weekly for up to an additional 6 months in the absence of unacceptable toxicity. Patients receive treatment at the same dose level as on protocol MSKCC-01131.

Patients are followed at approximately 30 days.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable relapsed or refractory solid tumor or non-Hodgkin's lymphoma that has been treated on MSKCC-01131
* Must have completed participation in protocol MSKCC-01131 through visit 16 and have shown evidence of stable disease or complete or partial remission of tumor burden and no evidence of symptomatic deterioration

  * No adverse event or toxicity which resulted in discontinuation of participation in protocol MSKCC-01131
  * If a patient experienced dose-limiting toxicity, then the patient must have demonstrated the ability to tolerate the same dose or a lower dose prior to entry in this study
* No known or suspected squamous cell carcinoma of the lung
* No prior or concurrent new neurological symptoms or CNS (brain or leptomeningeal) metastases during protocol MSKCC-01131

PATIENT CHARACTERISTICS:

Age

* 25 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 9.0 g/dL
* No severe or uncontrolled hematologic condition

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN
* Alkaline phosphatase no greater than 2 times ULN
* PT, PTT, and INR normal

Renal

* Creatinine no greater than ULN
* No 1+ or greater proteinuria
* No severe or uncontrolled renal condition

Cardiovascular

* No severe or uncontrolled cardiovascular condition

Pulmonary

* No severe or uncontrolled pulmonary condition

Other

* No prior hypersensitivity reactions to any recombinant proteins (e.g., VEGF Trap)
* No severe or uncontrolled gastrointestinal, immunological, or musculoskeletal condition
* No severe or uncontrolled psychiatric condition or adverse social circumstance that would preclude study
* No other condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent epoetin alfa, filgrastim (G-CSF), or sargramostim (GM-CSF)
* No other concurrent immunotherapy

Chemotherapy

* No concurrent standard chemotherapy

Endocrine therapy

* No concurrent adrenal corticosteroids except low doses as replacement therapy in patients who have previously received suppressive doses or for adrenal insufficiency
* No concurrent systemic hormonal contraceptive agents

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* At least 30 days since prior investigational therapy other than VEGF Trap
* No concurrent standard or other investigational anticancer agents
* No concurrent herbal supplements ("nutraceuticals")
* No concurrent anticoagulant or antiplatelet drugs (e.g., warfarin, heparin, aspirin, or other nonsteroidal anti-inflammatory drugs) except selective cyclo-oxygenase-2 (COX-2) inhibitors for analgesia
* No concurrent COX-2 inhibitors for tumor treatment or prophylaxis

Ages: 25 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Dupont, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Dupont J, Camastra D, Gordon MS, et al.: Phase 1 study of VEGF Trap in patients with solid tumors and lymphoma. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-776, 2003.
- [Result] Tew WP, Gordon M, Murren J, Dupont J, Pezzulli S, Aghajanian C, Sabbatini P, Mendelson D, Schwartz L, Gettinger S, Psyrri A, Cedarbaum JM, Spriggs DR. Phase 1 study of aflibercept administered subcutaneously to patients with advanced solid tumors. Clin Cancer Res. 2010 Jan 1;16(1):358-66. doi: 10.1158/1078-0432.CCR-09-2103. Epub 2009 Dec 22. PMID 20028764